CLINICAL TRIAL: NCT03096392
Title: A Randomized Controlled Comparison of Hepatic Directed Vesicle (HDV)-Insulin Lispro Versus Insulin Lispro Alone to Further Improve Glycemic Control in Type 1 Diabetes Mellitus Subjects With Good Glycemic Control
Brief Title: Comparison of Hepatic Directed Vesicle (HDV)-Insulin Lispro Versus Insulin Lispro to Further Improve Glycemic Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diasome Pharmaceuticals (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP 01-2017-01
Record Dates: First submitted 2017-03-01; First posted 2017-03-30 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Double blind, active comparator controlled (insulin lispro) to HDV insulin lispro, multiple dose safety, tolerability and efficacy study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, investigators, monitors, sponsor and sponsor representatives are blinded to the treatment group and treatment to patients are randomized. The group randomizing the subjects, the pharmacist preparing the drug, the party shipping the drug are unblinded but do not have contact with the blinded parties. An unblinded monitor will monitor any activities performed by unblinded parties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HDV insulin lispro 100 UNT/mL (Experimental): insulin lispro with 0.8 ml HDV added to a 10 ml vial of insulin lispro, injected subcutaneous before meals as needed. Study duration of 7 weeks (6 weeks of treatment)
  Interventions: Drug: HDV insulin lispro 100 UNT/ML
- insulin lispro 100 UNT/ML (Active Comparator): insulin lispro with 0.8 ml sterile water for injection added to a 10 ml vial of insulin lispro, injected subcutaneous before meals as needed. Study duration of 7 weeks (6 weeks of treatment)
  Interventions: Drug: Insulin Lispro 100 UNT/ML

INTERVENTIONS:
Drug: HDV insulin lispro 100 UNT/ML — HDV is the active excipient, added to insulin lispro. HDV binds to a portion of the insulin lispro.
  Other Names: Hepatic Directed Vesicle insulin lispro 100 UNT/ML
  Arms: HDV insulin lispro 100 UNT/mL
Drug: Insulin Lispro 100 UNT/ML — Sterile Water for Injection is added to the insulin lispro, to dilute the insulin lispro equal to the HDV insulin lispro
  Other Names: Humalog
  Arms: insulin lispro 100 UNT/ML

SUMMARY:
Multi-Center, double blind, active comparator controlled multiple dose safety, tolerability and efficacy study

DETAILED DESCRIPTION:
This is a double blind, active comparator controlled multiple dose safety, tolerability and efficacy study comparing HDV insulin lispro with insulin lispro in 40 Type 1 Diabetes Mellitus Subjects with Good Glycemic Control, with specific focus on time in range (70-180 mg/dL). Subjects will be screened and then monitored with one week of baseline CGM. They will then be randomized to one of two treatment groups: (A) six weeks of treatment with HDV-lispro (B) six weeks of treatment with insulin lispro diluted with sterile water alone.

All subjects will use insulin glargine or insulin degludec for basal insulin coverage throughout the trial. Fasting glucose goals will be 70-120 mg/dL, with recommendations for dosage adjustments made twice weekly according to a simple dosing algorithm based on mean fasting glucose values during the previous 3-4 days.

Subjects will receive standard diabetes education refresher training at the beginning of the trial, including review of insulin dose administration and titration, carbohydrate counting (or other dietary planning as deemed appropriate by the investigator), avoidance of hypoglycemia, and management of exercise and stress.

Post meal (60-90 min after start of meal) goals will be <140 mg/dL. A test meal study (standardized liquid test meal) to be conducted at the beginning of treatment (baseline study) and at the end of the six week treatment period (treatment comparison study). Subjects will also perform blinded continuous glucose monitoring during 4 weeks of study (i.e weeks 1,3,5 and 7 of study)

Throughout study, subjects will be asked to perform frequent self-monitoring of blood glucose (SMBG), at least 6 times per day (before and 60-90 minutes after each meal) during 3 or more days of each week. This will serve as data for therapeutic decision-making as well as for data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of age 18 to 65 years, inclusive. Females of child-bearing potential must use a standard and effective means of birth control for the duration of the study
2. T1DM ≥12 months
3. C-peptide <0.6 ng/mL (single retest allowed)
4. Treatment with rapid analog insulin for the previous 6 months and willing to use insulin vial and syringe to deliver rapid acting insulin during the study
5. Currently using either insulin glargine (U100 only) or insulin degludec for basal insulin therapy for at least 4 weeks prior to study
6. Not using insulin pump delivery systems during the previous 3 months
7. Familiarity with continuous glucose monitoring (CGM) technology; subjects need to be not currently using CGM; subjects will NOT use unblinded CGM during the treatment period of the trial
8. Willingness to use insulin lispro as the analog bolus insulin during the study period
9. BMI ≥18.0 kg/m2 and ≤35.0 kg/m2
10. 6.9%≤A1C≤7.9% (single retest allowed)

Exclusion Criteria:

1. Known or suspected allergy to any component of any of the study drugs in this trial.
2. A patient who has unstable proliferative retinopathy or maculopathy, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator
3. As judged by the investigator, clinically significant active disease of the gastrointestinal, cardiovascular (including a history of arrhythmia or conduction delays on ECG), hepatic, neurological, renal, genitourinary, or hematological systems, or uncontrolled hypertension (diastolic blood pressure ≥ 100 mmHg and/or systolic blood pressure ≥ 160 mmHg after 5 minutes in the supine position).
4. History of any illness or disease that in the opinion of the Investigator might confound the results of the trial or pose additional risk in administering the study drugs to the patient.
5. As judged by the Investigator, clinically significant findings in routine laboratory data
6. Use of drugs that may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia
7. Use of oral anti-diabetic or non-insulin anti-diabetic injection therapies (e.g. SGLT-2 inhibitors, pramlintide, GLP-1 agonists, etc.) during the 4 weeks prior to randomization
8. Current smokers; if a former smoker, no tobacco products (inhaled, oral or buccal) for the previous 3 months
9. Use of e-cigarettes or other nicotine-containing products for the previous 3 months
10. Current addiction to alcohol or substances of abuse as determined by the Investigator.
11. Pregnancy, breast-feeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, intra-uterine device [IUD], oral or injectable contraceptives, barrier methods or abstinence as per investigator discretion).
12. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation in this study
13. Symptomatic gastroparesis.
14. Receipt of any investigational drug within 4 weeks of Visit 2 in this study
15. Any condition (intrinsic or extrinsic) that in the judgment of the Investigator will interfere with trial participation or evaluation of data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
The amount of time, in minutes, glucose levels are within range (70-180 mg/dL) | 6 weeks
  evaluate continuous glucose monitoring (CGM) profiles during treatment with HDV insulin lispro versus insulin lispro alone, with specific focus on time in range (70-180 mg/dL)

SECONDARY OUTCOMES:
The number of events that blood glucose is equal to or less than 70 mg/dL | 6 weeks
  evaluate hypoglycemia frequency and severity during treatment with HDV insulin lispro versus insulin lispro alone
The number of events blood glucose is less than 54 mg/dL | 6 weeks
  evaluate hypoglycemia frequency and severity during treatment with HDV insulin lispro versus insulin lispro alone
Postprandial glucose levels in mg/dL following test meal challenge | 6 weeks
  evaluate glucose response to a standardized test meal challenge following six weeks of treatment with HDV insulin lispro versus insulin lispro alone
HbA1c levels in percentage (%) at beginning of trial compared to HbA1c levels at the end of the study | 6 weeks
  evaluate overall glycemic control (A1C) following six weeks of treatment with HDV insulin lispro versus insulin lispro alone
Self-Monitoring Blood Glucose (SMBG) results in mg/dL before and after every meal | 6 weeks
  evaluate self-monitoring of blood glucose (SMBG) values before and after meals during treatment with HDV insulin lispro versus insulin lispro alone
Total doses of insulin used (in number of units of insulin injected) during the study | 6 weeks
  compare insulin doses (prandial, basal and total) during HDV insulin lispro treatment versus insulin lispro alone

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B Muchmore, MD, Study Director — Chief Medical Officer
Locations (4):
- United States (4):
  - Barbara Davis Center for Diabetes, University of Colorado, Aurora, Colorado
  - Baptist Diabetes Associates, Miami, Florida
  - Lucas Research, Inc., Morehead City, North Carolina
  - Texas Diabetes and Endocrinology, Austin, Texas

IPD SHARING:
Plan to Share IPD: No
Not planned